CLINICAL TRIAL: NCT05814601
Title: Effect pf Preemptive Low Dose Norepinephrine Infusion on Hemodynamic Stability in Brain Tumor Resection
Brief Title: Effect of Preemptive Low Dose Norepinephrine Infusion on Intraoperative Hemodynamic Stability and Postoperative Outcomes in Patients Undergoing Brain Tumor Resection With a Craniotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4-2022-1619
Record Dates: First submitted 2023-02-28; First posted 2023-04-18 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms | interventions — Norepinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): norepinephrine at a concentration of 5 mcg/ml is preemptively administered
  Interventions: Drug: norepinephrine
- Control group (No Intervention): norepinephrine at a concentration of 5 mcg/ml is not preemptively administered

INTERVENTIONS:
Drug: norepinephrine — norepinephrine at a concentration of 5 mcg/ml is preemptively administered
  Arms: experimental group

SUMMARY:
In the experimental group, norepinephrine at a concentration of 5 mcg/ml is preemptively administered through peripheral venous catheter with a size of 20 G or more from the time of anesthesia induction to the end of anesthetic administration. The norepinephrine is not preemptively administered in the control group. For anesthesia, total intravenous anesthesia using propofol and remifentanil is performed. During anesthesia, the injection rate of the test drug is allowed to be adjusted according to the blood pressure within the permissible range, and anesthesia management such as fluid infusion, blood transfusions, and drug administration is performed according to the judgment of the anesthesiologist, and there are no restrictions.

The achievement of hemodynamic stability during anesthesia is judged by the percentage (%) of the time when the target blood pressure falls outside of 90-110%, 80-120%, and 70-130% of the target blood pressure during the total anesthesia duration. The number of hemodynamic unstability occurred, and the number of patients with hemodynamic unstability are also sought. The incidence of postoperative complications between the two groups is also compared.

ELIGIBILITY:
Inclusion Criteria:

Patients aged 20 to 65 who undergo elective craniotomy for brain tumor resection

Exclusion Criteria:

1. emergency surgery
2. If the subject includes those who cannot read the consent form (e.g. illiterate, foreigners, etc.)
3. cognitive dysfunction
4. pregnant, lactating
5. Congestive heart failure (New York Heart Association scores ≥3)
6. arrhythmia
7. Renal dysfunction (estimated Glomerular Filtration Rate less than 30 ml/min/1.73m2)
8. Patients with severe respiratory disease (pneumonia, chronic obstructive pulmonary disease, asthma under treatment, etc.)
9. Uncontrolled hypertension (baseline blood pressure greater than 140/90)

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
the percentage (%) of the time when the target blood pressure falls outside of 90-110%, 80-120%, and 70-130% of the target blood pressure during the total anesthesia duration | during the total anesthesia duration (maximum up to 24 hours)
The number of hemodynamic unstability occurred | during the total anesthesia duration (maximum up to 24 hours)
  ※ hemodynamic unstability is defined when the target blood pressure falls outside of 90-110%, 80-120%, and 70-130% of the target blood pressure
The number of patients with hemodynamic unstability | during the total anesthesia duration (maximum up to 24 hours)
  ※ hemodynamic unstability is defined when the target blood pressure falls outside of 90-110%, 80-120%, and 70-130% of the target blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Hye Jin Kim, Principal Investigator — Department of Anesthesiology and Pain Medicine, Yonsei University College of Medicine
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No